CLINICAL TRIAL: NCT03942523
Title: School-based Interventions to Promote Personal and Environmental Hygiene Among Children in Pakistan: Protocol for a Mixed Methods Study
Brief Title: Intervention to Promote Hygiene Behavior Among School Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Nousheen Pradhan, Senior Instructor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PF90/1016)
Record Dates: First submitted 2019-05-01; First posted 2019-05-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Behavioral Assessment of Children; Communicable Diseases in Children

STUDY DESIGN:
Intervention Model Description: Behavior change communication sessions will be administered to school children belonging to 1-5 grades in schools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School Children (Experimental): School children will be administered with behavioral change communication sessions as an intervention
  Interventions: Behavioral: Behavior Change Communication to promote hygiene behavior

INTERVENTIONS:
Behavioral: Behavior Change Communication to promote hygiene behavior — Behavior Change Communication sessions will be used to promote knowledge and practices among young children and to prevent communicable diseases.
  This will include, capacity building of teachers and students, health awareness sessions at the school and improving school physical environment

SUMMARY:
Background: Poor personal hygiene and inadequate sanitation practices among young children in Low Middle Income Countries such as Pakistan can lead to critical, life-threatening illnesses such as respiratory infections, diarrheal disease, malnutrition and developmental delays. An intervention for personal/environmental hygiene practices for primary schoolchildren will be implemented at schools in urban squatter settlements of Karachi, Pakistan, aiming to improve the hygiene knowledge and practices (K&P) amongst primary schoolchildren and their mothers (participants), while identifying facilitating and impeding factors in the adoption of hygiene practices for children.

Methods: The study will be built on quasi-experimental design with mixed methods data collection approaches. To assess primary grade children and their mothers' hygiene-status, K&P survey will be held in the pre-intervention phase. This phase also includes qualitative exploration of mothers' and teachers' perceptions about children's hygiene literacy, factors facilitating and impeding the adoption of the same among school children, for which in-depth guides and focus group discussion tools will be used with teachers and mothers respectively. School physical environmental assessment will be carried out pre-post intervention. This will be followed by multi-component intervention phase with behavior change strategies to improve children's and mothers' hygiene K&P. The post-intervention phase will assess the intervention effectiveness in terms of enhancing hygiene K&P among schoolchildren and mothers, alongside exploration of mothers and teachers' insights into whether or not the intervention has brought changes in improving hygiene practices among children.

Results: Paired T-test will be done pre-post intervention to measure the differences in knowledge and practice scores between mothers' hygiene literacy and practices with their child's knowledge and practices. Similar test will also be run to assess the differences in children' hygiene knowledge and practice scores pre and post intervention. Thematic analysis will be used for qualitative data.

Discussion: Multi-component intervention aimed at improving personal and environmental hygiene among primary school children offers an opportunity to design and test various behavioral change strategies at school and home setting. The study findings will be significant in assessing the intervention effectiveness in improving children's overall hygiene.

DETAILED DESCRIPTION:
Background:

Globally, communicable diseases are prevalent among school age children and the exposure to variety of pathogens causing preventable diseases in school population is inevitable. Underlying factors mainly rests on poor personal hygiene and inadequate sanitation practices leading to school absenteeism and life threatening illnesses among children (if continually neglected in the long run). The situation is worse in low and middle income countries due to inadequate health care facilities leading to compromised health status of school children.

Among communicable diseases, respiratory infections and diarrheal diseases are regarded as the deadliest killers of young children. Incidence of diarrheal disease in the initial years has been linked with impaired cognitive performance in the later childhood. In addition, in developing countries intestinal helminthic infection is a commonly cited problem among school-age children. Furthermore, oral health cavity infections are also commonly found in school going children worldwide. Frequent attacks of infection predispose young children to malnutrition and can form a vicious circle and retard children's physical and cognitive development. Moreover, the contextual factors such as poor socio-economic environment further deteriorate the health status of school children especially in low and middle income countries.

In the Pakistani context, alongside pneumonia and diarrhea worm infestation and scabies among school age children are the commonly reported health issues; manifesting poor personal hygiene. An evaluation study on water, sanitation and hygiene intervention on school child performance in two cities showed that almost 48% of government school children avoid going to school toilets due to poor sanitary condition. In local context, studies are mostly focused on oral hygiene assessment among children, showing satisfactory knowledge about using tooth paste. Comprehensive assessment about personal and environmental hygiene assessment among children, teachers and parents has remained a gap. Poor knowledge and practice of, and attitudes to personal hygiene have negative consequences on their long term development. This necessitates the designing and testing of school-based interventions aiming to improve hygiene behaviors among children, thereby minimizing their potential to capture preventable illnesses.

It is unfortunate that school health remains a neglected aspect of public health in Pakistan. In 2005, School Health Program was launched in 17 districts of the country by Ministry of Education, Pakistan in collaboration with United Nations Educational, Scientific and Cultural Organization (UNESCO). The program focused on various components including personal hygiene and environmental education but its impact was not determined . To the best of our knowledge, there is paucity of studies in Pakistan on school-based interventions to promote personal and environmental hygiene of school children, with child's parents and teachers' involvement. Towards designing school based programs, role of parents and teachers must be considered as they are the important role models for school going age children. And thus had detrimental effects in shaping children's overall health and hygiene behavior.

In this paper, Investigators present a study protocol using mixed-methods study design to be implemented in schools of a peri-urban community setting, Pakistan. The proposed study aims to improve the knowledge and practices of school children towards personal and environmental hygiene through school based intervention. To our knowledge, holistic assessment of hygiene among school children has not been studied in the local context. And the intervention to be implemented (with behavior change communication using adult to child and child to child approach, assessment of education curriculum on hygiene concepts) has never been studied before.

Primary research questions

1. Does school-based hygiene intervention facilitate improvement in knowledge and practices among primary school children studying in semi urban schools, Pakistan?
2. What are the enablers and barriers towards the adoption of personal and environmental hygiene practices by school children?

Secondary research questions Does improvement in knowledge and practices among the mothers of primary school children studying in semi-urban schools contributes to improved knowledge and practices of school children?

Methods Study design The study will employ a quasi-experimental design (pre-post intervention without control arm). The proposed study design is chosen as it will facilitate in evaluating school based interventions in the selected school settings without randomization. Similar to the randomized trials, quasi-experiments (community based trial) aims to demonstrate causality between an intervention and an outcome at the defined interval.

Study settings The study will be conducted in District Malir, Gaddap town in Karachi, Pakistan

Data collection methods The study is built on mixed method data collection approaches to gain insight of the hygiene literacy and practices among school children, teachers and child's mothers. Table 1 lists different data collection methods with its purpose and interval.

Study phases The study has been structured into 3 phases - pre-intervention, intervention and post-intervention.

ELIGIBILITY:
Inclusion criteria for Schools:

* Primary schools run by government or / NGO functional in District Malir, Gaddap town of Karachi

Exclusion Criteria for Schools:

* Consent not given by school administration.

Inclusion Criteria for Children:

* Students enrolled in primary grade (class 1-5)
* Informed consent given by either of the child's parents.
* After obtaining child's parents' consent, assent obtained from children.

Exclusion Criteria for Children:

* Assent not obtained from children

Inclusion criteria for Mothers:

* Mothers whose children are studying in grade 1-5 in selected/sample schools will be recruited.
* Mothers available at the time of data collection
* Mothers who gave consent

Exclusion Criteria for Mothers:

* Mothers who didn't meet the above eligibility criteria is excluded to participate.

Inclusion Criteria for Teachers:

* Teachers who are involved in teaching grade 1-5 students in the selected schools.
* Those who are available at the time of the study will be recruited after their informed consent.

Exclusion Criteria for Teachers:

* Those teachers who didn't give consent will be excluded.

Inclusion Criteria for Key Stakeholders:

* District Education Officers (DEO) and District Health Officer (DHOs) who currently hold the offices will be interviewed.
* Interviews with these respondents will only be held after obtaining their informed consent.

Exclusion Criteria for Key Stakeholders:

* Stakeholders who didn't provide consent will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Improved hygiene knowledge and practices among young children through survey tool | 3-4 months
  Changes in knowledge and practice of school children regarding hygiene will be assessed. There are no sub-scales used in the study. All knowledge and practice related responses will be measured as scores (pre-post intervention). Scores will be summed together. Less than 50 will be considered as poor, minimum and maximum score for rest of the categories are 50-75 will be considered as Good and 75-100 as Excellent. Higher values in each of the three categories will represent better outcomes for knowledge and practice.

SECONDARY OUTCOMES:
Change prevalence of communicable diseases among young children through structured questionnaire | 3-4 months
  This will include assessment of the change in the prevalence of communicable diseases (diarrhea, typhoid, pneumonia, oral health infections, scabies, hepatitis and mosquito borne infections) through structured questionnaire. Proportions of the children with these conditions will be used to report the change. No scales or sub-scales will be used. Proportions specific for each diseases will be averaged out pre-post intervention study.

CONTACTS AND LOCATIONS:
Overall Officials: Nousheen A Pradhan, MSc, Principal Investigator — Senior Instructor
Locations (1):
- Aga khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
At this stage, I intend to disseminate the study results with researchers.

REFERENCES:
- [Background] Vivas AP, Gelaye B, Aboset N, Kumie A, Berhane Y, Williams MA. Knowledge, attitudes and practices (KAP) of hygiene among school children in Angolela, Ethiopia. J Prev Med Hyg. 2010 Jun;51(2):73-9. PMID 21155409
- [Background] Niehaus MD, Moore SR, Patrick PD, Derr LL, Lorntz B, Lima AA, Guerrant RL. Early childhood diarrhea is associated with diminished cognitive function 4 to 7 years later in children in a northeast Brazilian shantytown. Am J Trop Med Hyg. 2002 May;66(5):590-3. doi: 10.4269/ajtmh.2002.66.590. PMID 12201596
- [Background] Oliveira D, Ferreira FS, Atouguia J, Fortes F, Guerra A, Centeno-Lima S. Infection by Intestinal Parasites, Stunting and Anemia in School-Aged Children from Southern Angola. PLoS One. 2015 Sep 15;10(9):e0137327. doi: 10.1371/journal.pone.0137327. eCollection 2015. PMID 26371758
- [Background] Sarkar M. Personal hygiene among primary school children living in a slum of Kolkata, India. J Prev Med Hyg. 2013 Sep;54(3):153-8. PMID 24783893
- [Background] Haque SE, Rahman M, Itsuko K, Mutahara M, Kayako S, Tsutsumi A, Islam MJ, Mostofa MG. Effect of a school-based oral health education in preventing untreated dental caries and increasing knowledge, attitude, and practices among adolescents in Bangladesh. BMC Oral Health. 2016 Mar 25;16:44. doi: 10.1186/s12903-016-0202-3. PMID 27016080
- [Background] Aiello AE, Coulborn RM, Perez V, Larson EL. Effect of hand hygiene on infectious disease risk in the community setting: a meta-analysis. Am J Public Health. 2008 Aug;98(8):1372-81. doi: 10.2105/AJPH.2007.124610. Epub 2008 Jun 12. PMID 18556606
- [Derived] Pradhan NA, Mughis W, Ali TS, Naseem M, Karmaliani R. School-based interventions to promote personal and environmental hygiene practices among children in Pakistan: protocol for a mixed methods study. BMC Public Health. 2020 Apr 14;20(1):481. doi: 10.1186/s12889-020-08511-0. PMID 32290822

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03942523/Prot_SAP_001.pdf